CLINICAL TRIAL: NCT06124417
Title: The Efficacy and Safety of Sertraline in Maintenance Hemodialysis Patients With Depression: a Randomized Controlled Study
Brief Title: Efficacy and Safety of Sertraline in the Treatment of Maintenance Hemodialysis Patients With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yunfeng Xia, Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The First Chongqing MU
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Efficacy, Team; Adverse Reaction to Drug
Keywords: Hemodialysis; Depression; Sertraline; Efficacy; Safety
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The Hamilton Rating Scale for Depression (HAMD) will be applied to assess the depressive status of all enrolled patients. This scale consists of 24 survey items, each with a score of 0-4. Patients will be assigned to the treatment group if their score was ≥8. Patients were given sertraline for antidepressant treatment in the treatment group. The initial dose ranged from 25 to 50 mg, taken orally once daily, and the dosage was adjusted based on the patient's response to the medication.
  Interventions: Drug: Sertraline
- Control group (No Intervention): Patients will be assigned to the control group if their HAMD score was <8.

INTERVENTIONS:
Drug: Sertraline — The initial dose ranged from 25 to 50 mg, taken orally once daily, and the dosage was adjusted based on the patient's response to the medication.
  Other Names: Conventional treatment
  Arms: Treatment group

SUMMARY:
Depression is a common mental disorder in patients undergoing maintenance hemodialysis (MHD), which increases the risk of cardiovascular events, hospitalization rates, and mortality, but has not received enough attention from patients and medical staff. Sertraline is a selective serotonin reuptake inhibitor with fewer adverse reactions and higher safety compared to other antidepressants. This study aims to investigate the efficacy and safety of sertraline in patients undergoing MHD with depression.

This study used a randomized controlled design and evaluated the depression status of the patients using the Hamilton Depression Scale (HAMD). MHD patients with comorbid depression were recruited and divided into the treatment group and the control group. The treatment group received sertraline for antidepressant therapy, while the control group did not receive any antidepressant medication. To investigate the efficacy and safety of sertraline before and after intervention.

DETAILED DESCRIPTION:
The HAMD, the Medication Adherence Report Scale-5 (MARS-5), the Mini Nutritional Assessment short-form (MNA-SF) and the Kidney Disease Quality of Life-36 (KDQOL-36) scales were used to evaluate changes in depression status, quality of life, medication adherence and nutritional status before and after the intervention. Clinical and laboratory indicators were collected before and after the intervention. Adverse reactions during the intervention were also recorded.

The initial dose ranged from 25 to 50 mg, taken orally once daily, and the dosage was adjusted based on the patient's response to the medication. In the control group, no antidepressant treatment was given.

ELIGIBILITY:
Inclusion Criteria:

1. Long-term MHD patients in the blood purification center of our hospital, older than 18 years old, maintenance dialysis for at least 3 months, 2-3 times a week, 3-4.5 hours each time;
2. Meet the CKD5 diagnostic criteria;
3. The cardiopulmonary function was relatively stable before enrollment, and the life expectancy was more than 1 year;
4. The clinical data were basically complete;
5. Consciousness, intelligence is normal, can understand the questionnaire content.

Exclusion Criteria:

1. Communication, communication disorders or other psychiatric history;
2. Combined with active pulmonary tuberculosis, AIDS, severe infection patients;
3. Pregnant or lactating women;
4. Those who are taking antidepressants or other antipsychotic drugs;
5. Unable or unwilling to cooperate with the researcher.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
HAMD score | 12 weeks
  If there is no decrease in HAMD score after treatment, it is considered ineffective. If the score decreases but remains ≥8, it is considered partial improvement. If the score decreases to below 8, it is considered complete remission.
KDQOL-36 score | 12 weeks
  If the KDQOL-36 score increases, the quality of life is considered to be improved.
Incidence of Adverse events reaction | 12 weeks
  Including nausea, diarrhea, constipation, anorexia, dry mouth, drowsiness, dizziness, and headache.

CONTACTS AND LOCATIONS:
Overall Officials: Yunfeng Xia, Dr., Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided